CLINICAL TRIAL: NCT05925764
Title: Whole Slide Image Based Deep Learning for Diagnosing the International Association for the Study of Lung Cancer Proposed Grading System of Lung Adenocarcinoma
Brief Title: WSI Based DL for Diagnosing the IASLC Grading System of Lung Adenocarcinoma
Status: Recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Chang Chen, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: WSIGS
Record Dates: First submitted 2023-05-12; First posted 2023-06-29 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Lung Adenocarcinoma; Whole Slide Image; IASLC Grading System; Artificial Intelligence
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Whole Slide Image based Deep Learning — Whole Slide Image Based Deep Learning for Diagnosing the IASLC Grading System of Lung Adenocarcinoma

SUMMARY:
The purpose of this study is to evaluate the performance of a whole slide image based deep learning model for diagnosing the IASLC grading system in resected lung adenocarcinoma based on a multicenter prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age ranging from 18-85 years old;
2. Pathological confirmation of primary lung adenocarcinoma after surgery;
3. Obtained written informed consent.

Exclusion Criteria:

1. Multiple lung lesions;
2. Poor quality of whole slide images;
3. Mucinous adenocarcinomas and variants;
4. Participants who have received neoadjuvant therapy.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Resected Lung Adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Agreement rate of the IASLC grading system | 2024.11.01-2024.12.31
  Agreement rate between the deep learning model and pathologists in diagnosing the IASLC grade of lung adenocarcinoma.

SECONDARY OUTCOMES:
Agreement rate of the predominant subtypes | 2024.11.01-2024.12.31
  Agreement rate between the deep learning model and pathologists in diagnosing the predominant growth patterns of lung adenocarcinoma.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Ningbo HwaMei Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: No